CLINICAL TRIAL: NCT01592669
Title: The Effect of Passive Leg Raising or Experimental Clinical Practices on the Prevention of Hypotension Following Tourniquet Release in Total Knee Arthroplasty Patients
Brief Title: Passive Leg Raising Attenuates and Delays Tourniquet Deflation-induced Hypotension and Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Go-Shine Huang, Clinical assistant professor. Doctor of anesthesiology and critical care, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TSGH-C101-105
Record Dates: First submitted 2012-03-30; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Hypotension; Tachycardia
Keywords: Passive leg raising, blood pressure, heart rate
MeSH Terms: conditions — Hypotension; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- passive leg group (Experimental): bilateral PLR was achieved by raising the patient's legs to a 45 angle.
  Interventions: Procedure: passive leg raising
- control (No Intervention): supine baseline position

INTERVENTIONS:
Procedure: passive leg raising — bilateral PLR was achieved by raising the legs of patient
  Other Names: PLR
  Arms: passive leg group

SUMMARY:
Background:

The pneumatic tourniquet is frequently used in total knee arthroplasty. Tourniquet deflation may result in hypotension and tachycardia caused by the rapid shift of blood volume back to the ischemic limb and a decrease in cardiac preload. Passive leg raising (PLR) represents a "self-volume challenge" that can result in an increase in preload. Such a PLR-induced increase in preload was hypothesized to attenuate the decrease in preload resulting from tourniquet deflation. This study was designed to evaluate the effect of PLR on hypotension and tachycardia following tourniquet deflation.

Methods:

Seventy patients who underwent unilateral total knee arthroplasty were assigned to either the bilateral PLR group (n = 35) or the control group (n = 35), in a prospective randomized trial. The patients' blood pressure and heart rate were measured before, during, and after tourniquet deflation.

DETAILED DESCRIPTION:
This study was a prospective randomized trial, which was approved by the Institutional Review Board of the hospital, and informed consent was obtained from each patient enrolled in the study. Patients with degenerative joint disease of the knee scheduled to receive unilateral total knee arthroplasty were enrolled in this study within one year. Exclusion criteria were bilateral total knee arthroplasty, previous knee surgery, cardiac arrhythmia, uncontrolled hypertension (systolic blood pressure > 170 mmHg), presence of a known aortic aneurysm, recent stroke or myocardial infarction, unstable angina pectoris, New York Heart Association functional class III or IV, and American Society of Anesthesiologists physical status IV to V. A series of numbered, opaque, sealed envelopes were used to randomly allocate participants to the bilateral PLR group (n = 35) or to the control group (n = 35). The trial flow chart is illustrated in Figure 1. The primary outcome measures were the blood pressure and heart rate before, during, and after tourniquet deflation.

The sample size estimate, based on previous studies8, indicated that 35 patients were required for each group in order to have a 90% chance of detecting a significant difference (P = 0.05, two-sided) between the groups. Patients were premedicated with fentanyl and/or midazolam for anxiolysis 5 min before induction of anesthesia. Spinal anesthesia was performed via the L3-L4 or L4-L5 interspace with a single dose of isobaric bupivacaine. A drop in systolic blood pressure to lower than 90 mmHg triggered ephedrine administration during the study.

Figure 2 illustrates the study protocol, which was divided into 4 steps. Blood pressure and heart rate were measured at each time point (T1-T17) throughout the protocol. Systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean blood pressure (MBP) were measured using noninvasive, automated techniques and a continuous electrocardiogram allowed measurements of heart rate. In addition, the doses of bupivacaine and ephedrine administrated, as well as the upper anesthetized level, and total fluid volume administered before tourniquet deflation were recorded.

Step 1 (T1-T5): In both groups, after induction of spinal anesthesia, the patient was placed in a supine position with a well-padded proximal tourniquet. The leg was exsanguinated with an Esmarch bandage, and a pneumatic tourniquet was applied and inflated to a pressure of 280-300 mm Hg, followed by the arthroplastic surgery. Recordings and measurements were taken at 30, 15, 10, 5, and 1 min before bilateral PLR (step 2).

Step 2 (T6-T7): In the PLR group, at the completion of the total knee arthroplasty, bilateral PLR was achieved by raising the patient's legs to a 45 degree angle. Recordings and measurements were taken 2 and 4 min after initiation of PLR. In the control patients, the legs were left in the baseline position, but hemodynamic measurements were still taken at time points corresponding to those in the PLR group.

Step 3 (T8-T10): In the PLR group, PLR was maintained and the tourniquet was deflated and hemodynamic recordings and measurements were taken at 2, 4, and 6 min after tourniquet deflation. At this step, blood pressure and heart rate were recorded for 6 min because previous reports have suggested that the nadir of the blood pressure occurred within 5 min after tourniquet deflation. In the control group, the tourniquet was deflated while the patient's legs remained in the baseline position and hemodynamic measurements were obtained at points corresponding to those in the PLR patients.

Step 4 (T11-T17): In the PLR group, the legs were returned to the baseline position and a fourth set of recordings and hemodynamic measurements were obtained 1, 3, 5, 10, 15, 30, and 60 min later. In the control group, the legs remained in the baseline position and corresponding hemodynamic measurements were obtained.

Statistical Methods Differences in demographic characteristics and perioperative data between the PLR and control patients were examined using chi-square or Student's t tests, depending on the measure. Hemodynamic measurements were analyzed over time by comparing the T6-T17 measurements to the T5 measurements in each group. Intragroup hemodynamic changes were analyzed using repeated measures one-way analysis of variance, followed by the Fisher's least-significant difference post-test. The generalized estimating equations test was used to compare the differences between groups (PLR and control group), with respect to blood pressure and heart rate measurements. The difference in the length of time from tourniquet deflation to the nadir in blood pressure between the groups was determined by Student's t test. The SPSS software (Version 15 SPSS Inc., Chicago, Illinois) was used for all analyses. All the tests were two-sided, and P < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative joint disease of the knee scheduled to receive unilateral total knee arthroplasty

Exclusion Criteria:

* bilateral total knee arthroplasty, previous knee surgery, cardiac arrhythmia, uncontrolled hypertension (systolic blood pressure > 170 mmHg), presence of a known aortic aneurysm, recent stroke or myocardial infarction, unstable angina pectoris, New York Heart Association functional class III or IV, and American Society of Anesthesiologists physical status IV to V

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Blood pressure | Baseline and 60 min
  The patients' blood pressure was measured before, during, and after tourniquet deflation. Step 1 (T1-T5), measurements were taken at 30, 15, 10, 5, and 1 min before bilateral passive leg raising (PLR). Step 2 (T6-T7), measurements were taken 2 and 4 min after initiation of PLR. Step 3 (T8-T10), measurements were taken at 2, 4, and 6 min after tourniquet deflation. Step 4 (T11-T17), measurements were obtained 1, 3, 5, 10, 15, 30, and 60 min later. Hemodynamic measurements and change were analyzed over time by comparing the T6-T17 measurements to the T5 measurements in each group.

SECONDARY OUTCOMES:
Heart rate | up to 60 min
  The patients' heart rate was measured before, during, and after tourniquet deflation. Step 1 (T1-T5), measurements were taken at 30, 15, 10, 5, and 1 min before bilateral passive leg raising (PLR). Step 2 (T6-T7), measurements were taken 2 and 4 min after initiation of PLR. Step 3 (T8-T10), measurements were taken at 2, 4, and 6 min after tourniquet deflation. Step 4 (T11-T17), measurements were obtained 1, 3, 5, 10, 15, 30, and 60 min later.Hemodynamic measurements and change were analyzed over time by comparing the T6-T17 measurements to the T5 measurements in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Go-shine Huang, MD, Principal Investigator — Department of Anesthesiology, Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Nei-Hu, Taipei, Taiwan

REFERENCES:
- [Derived] Huang GS, Wang CC, Hu MH, Cherng CH, Lee MS, Tsai CS, Chan WH, Hsieh XX, Lin LC. Bilateral passive leg raising attenuates and delays tourniquet deflation-induced hypotension and tachycardia under spinal anaesthesia: a randomised controlled trial. Eur J Anaesthesiol. 2014 Jan;31(1):15-22. doi: 10.1097/EJA.0b013e32836286e3. PMID 23812622